CLINICAL TRIAL: NCT02638831
Title: Open Label Randomized Study for Evaluating Efficacy and Safety of Ketorolac Tromethamine and Ketoprofen in Gel in Patients With Gonarthrosis and Low Back Pain
Brief Title: Ketorol Gel in Gonarthrosis and Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRL_RUS/PMS/2012/KETG
Record Dates: First submitted 2015-12-01; First posted 2015-12-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Gonarthrosis; Low Back Pain
Keywords: Pain; Gonarthrosis; Low Back Pain; Ketorolac Tromethamine; Ketoprofen
MeSH Terms: conditions — Osteoarthritis, Knee; Low Back Pain; Pain | interventions — Ketorolac Tromethamine; Ketoprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac Tromethamine (Experimental): Ketorolac 2% for external application. Column of gel about 3-5 cm is applied on the area of maximum pain three times a day for 10 days
  Interventions: Drug: Ketorolac Tromethamine
- Ketoprofen (Active Comparator): Ketoprofen gel 2.5% for external application. Column of gel (3-5 cm) is applied with a thin layer on the skin in the area of maximum pain 3 times a day for 10 days
  Interventions: Drug: Ketoprofen

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Ketorolac tromethamine gel 2% for external application. Column of gel about 3-5 cm is applied on the area of maximum pain three times a day for 10 days
  Arms: Ketorolac Tromethamine
Drug: Ketoprofen — Ketoprofen gel 2.5% for external application Column of gel (3-5 cm) is applied with a thin layer on the skin in the area of maximum pain 3 times a day for 10 days
  Arms: Ketoprofen

SUMMARY:
Comparative clinical study of Ketorolac tromethamineand Ketoprofen gel in patients with Gonarthrosis and Low back pain.

DETAILED DESCRIPTION:
This is a Comparative evaluation of therapeutic efficacy and safety of use of drug Ketorolac tromethamine gel and drug Ketoprofen gel , as an agent of local symptomatic therapy in patients with diseases of musculoskeletal system with associated pain syndrome in outpatient conditions.

The study includes patients with moderate pain syndrome in gonarthrosis and lower back pain (LBP).

The sample size of 240 was calculated for the main efficacy variable - mean pain intensity according to the visual analogue scale (VAS) in 10 days of therapy.

Patients who subjected to inclusion into the study and had signed informed consent will be distributed into the study groups depending on established diagnosis: Gonarthrosis group and LBP group.

ELIGIBILITY:
General inclusion criteria:

1. Patients of both sexes in the age group from 20 to 70 years, who have signed informed consent for participation in the study.
2. Understanding of spoken or written communication, adequate for being able to follow procedures of the Protocol and fill in documents related to the study.
3. For women: patients who are not pregnant, not breast-feeding. The female patients must be in either the post-climacteric period or surgically sterile, or for the entire period of the study use contraceptive methods with a reliability level of higher than 90%. Methods of contraception with higher than 90% level of reliability of common use include cervical caps with spermicide, diaphragms with spermicide, condoms, oral contraceptives.

Criteria of inclusion in the group "gonarthrosis":

1. Patients of both sexes in the age group from 40 to 70 years.
2. Roentgenologically confirmed gonarthrosis (presence of roentgenological symptoms of osteophytes and stenosis of joint space).
3. Intensity of pain in the knee joint as per visual analogue scale (VAS), when still: ≥40 mm, during movement: ≥ 50 mm.
4. Presence of one of the under mentioned combinations of criteria:

   1. Pain in the knee joint during the last one month, accompanied by crepitation in active movement of the joint, morning stiffness up to 30 min, age - 38 years and older.
   2. Pain in the knee joint during the last one month, accompanied by crepitation in active movement of the joint, morning stiffness up to 30 min., bone enlargements in the joint area.
   3. Pain in knee joint during the last one month in the absence of crepitation, bone enlargements in joint area

   Criteria of inclusion in the group "low backpain" :
5. Patients of both sexes in the age group of 20 to 65 years with acute pain syndrome in the lower part of the back (less than 12 weeks).
6. Intensity of pain in the back as per VAS when still ≥40 mm, during movement ≥ 50 mm.

Exclusion Criteria:

* 1. Feedback on Informed Consent Form signed by the patient for participation in the Study.

  2. Continuation of participation in the study is in conflict with the patient's interests.

  3. Occurrence of a serious adverse event in the patient, the relation of which to the administration of the drug under study is classified definite, probable or possible.

  4. Patient needs additional treatment which may affect the parameters of efficacy under study.

  5. Violations of the protocol, which in the opinion of the investigator or sponsor of the study, are significant for evaluation of results of the clinical trial.

  6. Discontinuation of the study by the sponsor. 7. Discontinuation of the study by the investigator. 8. Discontinuation of the study by the regulatory bodies.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in pain on visual analogue scale (VAS) from baseline | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Nadezhda A Shostak, PhD, Principal Investigator — 1 Russian National Research Medical Institute State Budgetary Institution of Higher Professional Education "N.I. Pirogov Russian National Research Medical Institute" of the Ministry of Health of Russia